CLINICAL TRIAL: NCT02539134
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Multiple Doses of TAK-935 in Healthy Subjects
Brief Title: TAK-935 Multiple Rising Dose Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-935-1002; U1111-1168-6634 (Registry Identifier: WHO)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-04

CONDITIONS: Epilepsy
Keywords: Drug therapy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1, Cohort 1: TAK-935 100 mg QD (Experimental): TAK-935 100 milligram (mg), solution, orally, once daily (QD) or TAK-935 placebo-matching solution, orally, QD for up to 14 days.
  Interventions: Drug: TAK-935; Drug: Placebo
- Part 1, Cohort 2: TAK-935 300 mg QD (Experimental): TAK-935 300 mg, solution, orally, QD or TAK-935 placebo-matching solution, orally, QD for up to 14 days.
  Interventions: Drug: TAK-935; Drug: Placebo
- Part 1, Cohort 3: TAK-935 300 mg BID (Experimental): TAK-935 300 mg, solution, orally, twice daily (BID) or TAK-935 placebo-matching solution, orally, BID for up to 10 days.
  Interventions: Drug: TAK-935; Drug: Placebo
- Part 1, Cohort 4: TAK-935 600 mg QD (Experimental): TAK-935 600 mg, solution, orally, QD or TAK-935 placebo-matching solution, orally, QD for up to 10 days.
  Interventions: Drug: TAK-935; Drug: Placebo
- Part 1, Cohort 5: TAK-935 400 mg QD (Experimental): TAK-935 400 mg, solution, orally, QD or TAK-935 placebo-matching solution, orally, QD for up to 14 days.
  Interventions: Drug: TAK-935; Drug: Placebo
- Part 2, Cohort 6: TAK-935 Dose 1 (Experimental): TAK-935 first decided dose as determined from other TAK-935 trials and Cohorts 1 to 4 of Part 1, solution, orally, QD or TAK-935 placebo-matching solution, orally, QD for up to 14 days.
  Interventions: Drug: TAK-935; Drug: Placebo
- Part 2, Cohort 7: TAK-935 Dose 2 (Experimental): TAK-935 second decided dose as determined from other TAK-935 trials and Cohorts 1 to 4 of Part 1, solution, orally, QD or TAK-935 placebo-matching solution, orally, QD for up to 14 days.
  Interventions: Drug: TAK-935; Drug: Placebo

INTERVENTIONS:
Drug: TAK-935 — TAK-935 oral solution
Drug: Placebo — TAK-935 placebo-matching oral solution

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of multiple rising doses of TAK-935 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935. This study will look at the pharmacokinetics, safety and tolerability of TAK-935 in healthy participants. The study will enroll approximately 56 participants. Participants will be randomly assigned (by chance, like flipping a coin) to 1 of the 5 cohorts in Part 1, which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Part 1, Cohort 1: TAK-935 100 mg QD
* Part 1, Cohort 2: TAK-935 300 mg QD
* Part 1, Cohort 3: TAK-935 300 mg BID
* Part 1, Cohort 4: TAK-935 600 mg QD
* Part 1, Cohort 5: TAK-935 400 mg QD Participants will be asked to take the oral solution once or twice a day at the same time for 14 days. An optional Part 2 may be conducted for collecting data to assess the engagement by TAK-935 of the central molecular target cholesterol 24S-hydroxylase (CH24H) by measuring the changes of levels of the metabolite 24S-hydroxycholesterol (24HC). In Part 2, participants will be assigned to up to 2 treatment groups at doses based on the data from other ongoing TAK-935 trials, combined with the safety and tolerability data from Cohorts 1-4 of Part 1.

This single center trial will be conducted in the United States. The overall time to participate in this study will be approximately 30 days. Participants will be admitted in the clinic for the first 14 days, and will be contacted by telephone on Day 28 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts

1. Is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy male or female aged 18 to 55 years inclusive, at the time of informed consent and first study medication dose.
4. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening and Day -1.
5. Male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
6. Female participant of childbearing potential who is sexually active with a non-sterilized male partner agrees to use routinely adequate contraception from signing of informed consent and throughout the duration of the study, and for 30 days after the last dose.
7. Can complete the CogState Battery at Screening.

   Additional Inclusion Criteria for Participants undergoing cerebrospinal fluid (CSF) Sampling (Part 2 only):
8. Agrees to spinal tap procedures for CSF collection.

Exclusion Criteria:

All Cohorts

1. Has received any investigational compound within 30 days prior to randomization.
2. Has received TAK-935 in a previous clinical study or as a therapeutic agent.
3. Has a significant history of uncontrolled, clinically significant neurologic (including seizure disorders), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease or psychiatric disorder or endocrine disease or other abnormality or any significant results from physical examinations, or clinical laboratory results which may impact the ability of the participant to participate or potentially confound the study results. It is the responsibility of the investigator to assess the clinical significance; however, consultation with the Takeda Medical Monitor may be warranted.
4. Has a known hypersensitivity to any component of the formulation of TAK-935.
5. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or a single measure of spirits or 1 small glass of wine.
6. Has taken any excluded medication, supplements, or food products during the time periods listed in the Excluded Medications and Dietary Products table.

   Additional Exclusion Criteria for Participants undergoing CSF sampling (Part 2)
7. Has CSF collection performed within 30 days prior to check-in (Day -3).
8. Has a known hypersensitivity to the anesthetic or its derivatives used during CSF collection, or any medication used to prepare the area of lumbar puncture.
9. Has significant vertebral deformities (scoliosis or kyphosis) which, in the opinion of the investigator, may interfere with lumbar puncture procedure.
10. Has a history of clinically significant back pain and/or injury.
11. Has local infection at the puncture site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 02 September 2015 to 19 April 2016.
Pre-assignment Details: Healthy participants received TAK-935 or placebo in Cohorts 1-5: 100 milligram(mg) once daily(QD), 300mg QD, 300mg twice daily(BID), 600mg QD, and 400mg QD respectively in Part 1. Study Part 2 (optional) was not conducted after review of initial data of TAK-935-1003(NCT02497235) along with safety and tolerability data from Cohorts 1 to 4 of Part 1.
Groups:
- Cohorts 1-5: Placebo: TAK-935 placebo-matching solution, orally, QD for up to 14 days in Cohorts 1, 2, and 5; BID for up to 10 days in Cohort 3 and QD for up to 10 days in Cohort 4.
- Cohort 1: TAK-935 100 mg QD: TAK-935 100 mg, solution, orally, QD for up to 14 days in Cohort 1.
- Cohort 2: TAK-935 300 mg QD: TAK-935 300 mg, solution, orally, QD for up to 14 days in Cohort 2.
- Cohort 3: TAK-935 300 mg BID: TAK-935 300 mg, solution, orally, BID for up to 10 days in Cohort 3.
- Cohort 5: TAK-935 400 mg QD: TAK-935 400 mg, solution, orally, QD for up to 14 days in Cohort 5.
- Cohort 4: TAK-935 600 mg QD: TAK-935 600 mg, solution, orally, QD for up to 10 days in Cohort 4.
Period: Overall Study
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Started | 10 | 6 | 6 | 6 | 6 | 6
Completed | 9 | 6 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (8.51) | 33.8 (4.62) | 33.7 (10.71) | 26.7 (4.50) | 37.7 (13.08) | 40.3 (11.55) | 34.5 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 2 | 0 | 10
  Male | 7 | 5 | 3 | 5 | 4 | 6 | 30
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 40
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 5 | 0 | 4 | 4 | 5 | 1 | 19
  Not Hispanic or Latino | 5 | 6 | 2 | 2 | 1 | 5 | 21
Race [Number; unit: participants]
  Black or African American | 3 | 1 | 2 | 1 | 1 | 1 | 9
  White | 7 | 5 | 4 | 5 | 5 | 5 | 31
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.7 (10.02) | 175.5 (5.65) | 165.5 (6.16) | 174.8 (8.57) | 167.5 (7.29) | 175.7 (5.43) | 172.0 (8.19)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 78.90 (13.136) | 79.37 (8.596) | 67.68 (10.860) | 73.55 (6.227) | 75.28 (12.367) | 78.25 (7.936) | 75.85 (10.647)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.30 (2.756) | 25.76 (2.386) | 24.66 (3.476) | 24.16 (2.629) | 26.67 (2.971) | 25.31 (1.491) | 25.56 (2.666)
Smoking Classification [Number; unit: participants]
  Never smoked | 7 | 5 | 6 | 6 | 4 | 4 | 32
  Ex-smoker | 3 | 1 | 0 | 0 | 2 | 2 | 8
Alcohol Classification [Number; unit: participants]
  Never drunk | 7 | 4 | 4 | 4 | 3 | 3 | 25
  Current drinker | 0 | 1 | 1 | 1 | 1 | 2 | 6
  Ex-drinker | 3 | 1 | 1 | 1 | 2 | 1 | 9
Xanthine/Caffeine Consumption [Number; unit: participants]
  Xanthine/Caffeine consumption | 6 | 2 | 4 | 2 | 3 | 4 | 21
  No Xanthine/Caffeine consumption | 4 | 4 | 2 | 4 | 3 | 2 | 19
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Female of childbearing potential | 2 | 1 | 3 | 1 | 1 | 0 | 8
  Not applicable (Male participant) | 7 | 5 | 3 | 5 | 4 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Day 1 up to Day 28
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 40.0 | 0 | 16.7 | 83.3 | 83.3 | 50.0

2. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Time Frame: Baseline up to Day 15
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 16.7 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Time Frame: Baseline up to Day 15
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 70 | 33.3 | 33.3 | 0 | 33.3 | 33.3

4. Primary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Safety 12-lead Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: Baseline up to Day 15
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 70.0 | 66.7 | 33.3 | 66.7 | 50.0 | 66.7

5. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-935
Time Frame: Day 1 and Day 14: Pre-dose and at multiple time points (up to 24 hours for Cohorts 1, 2, 4, and 5; up to 12 hours for Cohort 3) post-dose
Population: The pharmacokinetic (PK) set included all participants in the safety set who had at least 1 measurable plasma or urine concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  Day 1 | 418.536 (50.0) | 1729.173 (61.7) | 1269.337 (32.5) | 2374.498 (50.6) | 2448.500 (70.2)
  Day 14 | 469.137 (25.3) | 2865.655 (41.1) | NA (NA) — PK data for Cohort 3 was not available because dosing was discontinued on Day 10. | 2708.655 (40.3) | NA (NA) — PK data for Cohort 4 was not available because dosing was discontinued on Day 10.
Statistical Analysis 1: Comparison: Cohort 1: TAK-935 100 mg QD vs Cohort 2: TAK-935 300 mg QD vs Cohort 5: TAK-935 400 mg QD vs Cohort 4: TAK-935 600 mg QD; Day 1: For groups with QD dosing, dose proportionality for TAK-935 plasma exposure on Day 1 was assessed using the power model. For Day 1, the criteria for dose proportionality was the 90 percent (%) confidence interval (CI) for the slope within (0.875, 1.125) for the dose range of 100 mg to 600 mg; Test type: Superiority or Other; p = 0.757, Power model; Slope = 1.06, 90% CI 2-sided [0.741 to 1.374]
Statistical Analysis 2: Comparison: Cohort 1: TAK-935 100 mg QD vs Cohort 2: TAK-935 300 mg QD vs Cohort 5: TAK-935 400 mg QD; Day 14: For groups with QD dosing, dose proportionality for TAK-935 plasma exposure on Day 14 was assessed using the power model. For Day 14, the criteria for dose proportionality was the 90% CI for the slope within (0.839, 1.161) for the dose range of 100 mg to 400 mg; Test type: Superiority or Other; p = 0.042, Power model; Slope = 1.37, 90% CI 2-sided [1.078 to 1.664]

6. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-935
Time Frame: as for outcome 5
Population: The PK set included all participants in the safety set who had at least 1 measurable plasma or urine concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL)
  Day 1 | 423.284 (29.8) | 1794.084 (55.7) | 1250.256 (38.5) | 2281.664 (48.8) | 3563.187 (59.7)
  Day 14 | 435.232 (29.5) | 2494.972 (40.0) | NA (NA) — PK data for Cohort 3 was not available because dosing was discontinued on Day 10. | 2601.519 (40.4) | NA (NA) — PK data for Cohort 4 was not available because dosing was discontinued on Day 10.
Statistical Analysis 1: Comparison: Cohort 1: TAK-935 100 mg QD vs Cohort 2: TAK-935 300 mg QD vs Cohort 5: TAK-935 400 mg QD vs Cohort 4: TAK-935 600 mg QD; Day 1: For groups with QD dosing, dose proportionality for TAK-935 plasma exposure on Day 1 was assessed using the power model. For Day 1, the criteria for dose proportionality was the 90% CI for the slope within (0.875, 1.125) for the dose range of 100 mg to 600 mg; Test type: Superiority or Other; p = 0.191, Power model; Slope = 1.20, 90% CI 2-sided [0.946 to 1.450]
Statistical Analysis 2: Comparison: Cohort 1: TAK-935 100 mg QD vs Cohort 2: TAK-935 300 mg QD vs Cohort 5: TAK-935 400 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.036, Power model; Slope = 1.37, 90% CI 2-sided [1.089 to 1.657]

7. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-935
Time Frame: Day 1: Pre-dose and at multiple time points (up to 24 hours for Cohorts 1, 2, 4, and 5; up to 12 hours for Cohort 3) post-dose
Population: The PK set where Day 1 assessment for AUC∞ was available. The PK set included all participants in the safety set who had at least 1 measurable plasma or urine concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 6
ng*hr/mL | 427.418 (36.7) | 1811.936 (55.3) | 1397.108 (48.0) | 2310.461 (48.1) | 3606.449 (59.4)
Statistical Analysis 1: Comparison: Cohort 1: TAK-935 100 mg QD vs Cohort 2: TAK-935 300 mg QD vs Cohort 5: TAK-935 400 mg QD vs Cohort 4: TAK-935 600 mg QD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.288, Power model; Slope = 1.19, 90% CI 2-sided [0.890 to 1.489]

8. Secondary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Over the Dosing Interval for TAK-935
Time Frame: Day 14: Pre-dose and at multiple time points (up to 24 hours for Cohorts 1, 2, 4, and 5; up to 12 hours for Cohort 3) post-dose
Population: The PK set included all participants in the safety set who had at least 1 measurable plasma or urine concentration. No data was reported for Cohorts 3 and 4 since dosing was discontinued after Day 10.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Number analyzed (Participants) | 6 | 6 | 0 | 6 | 0
ng*hr/mL | 442.606 (28.4) | 2496.596 (40.0) |  | 2605.230 (40.3) |
Statistical Analysis 1: Comparison: Cohort 1: TAK-935 100 mg QD vs Cohort 2: TAK-935 300 mg QD vs Cohort 5: TAK-935 400 mg QD; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.039, Power model; Slope = 1.36, 90% CI 2-sided [1.080 to 1.642]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days after the last dose of double-blind study drug (Day 28)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-935 100 mg QD | Cohort 2: TAK-935 300 mg QD | Cohort 3: TAK-935 300 mg BID | Cohort 5: TAK-935 400 mg QD | Cohort 4: TAK-935 600 mg QD
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/10 | 0/6 | 1/6 | 5/6 | 5/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-5: Placebo (N=10) | Cohort 1: TAK-935 100 mg QD (N=6) | Cohort 2: TAK-935 300 mg QD (N=6) | Cohort 3: TAK-935 300 mg BID (N=6) | Cohort 5: TAK-935 400 mg QD (N=6) | Cohort 4: TAK-935 600 mg QD (N=6)
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Application site irritation (General disorders) | 3 | 0 | 1 | 0 | 2 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling of relaxation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Agraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual perseveration (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypervigilance (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Distractibility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tachyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.